CLINICAL TRIAL: NCT06542250
Title: A Modular Phase I/II Open-label Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD5492, a T Cell-engaging Antibody Targeting CD20 in Subjects With Relapsed or Refractory B-Cell Malignancies (TITANium)
Brief Title: A Study to Evaluate Safety, PK, PD and Efficacy of AZD5492, a T Cell-engaging Antibody Targeting CD20 in Subjects With R/R B-Cell Malignancies.
Acronym: TITANium
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9960C00001
Record Dates: First submitted 2024-07-29; First posted 2024-08-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: B-cell Malignancies
Keywords: CD20; CD8; T cell engager; TCR; AZD5492; Relapsed, Refractory; B-cell malignancies; CLL, Chronic lymphocytic leukemia; SLL, Small lymphocytic lymphoma; MCL, Mantle cell lymphoma; LBCL, Large B-cell lymphoma; FL, Follicular lymphoma; TITANium; TCE
MeSH Terms: conditions — Recurrence; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules each evaluating the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary efficacy of AZD5492 as monotherapy or in combination with other anticancer treatments in participants with R/R B-cell malignancies.
  - Module 1: AZD5492 Monotherapy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Module 1: AZD5492 Monotherapy (Experimental): AZD5492 monotherapy for Relapsed or Refractory B-Cell Malignancies.
  Interventions: Drug: AZD5492

INTERVENTIONS:
Drug: AZD5492 — CD8/TCR based T-cell engaging antibody targeting CD20, which is administered subcutaneously

SUMMARY:
This is a Phase I/II study designed to evaluate if experimental T cell engaging antibody targeting CD20 AZD5492 is safe, tolerable and efficacious in participants with Relapsed or Refractory B-Cell Malignancies.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Histologically documented CD20+ mature B-cell neoplasm

  * Large B-cell lymphoma
  * Follicular lymphoma
  * Mantle cell lymphoma
  * Chronic lymphocytic leukemia
  * Small lymphocytic lymphoma
* Relapsed, progressive and/or refractory disease following at least 2 prior lines of therapy;
* ECOG performance status of ≤ 2 (< 2 in EU countries).

The above is a summary, other inclusion criteria details may apply.

Exclusion Criteria:

* Any neoplasm histology not specified in the IC section;
* Active CNS involvement in lymphoma;
* CNS pathology including but not limited to any history of seizure disorder/epilepsy;
* Prior allogeneic HSCT within 180 days, prior autologous HSCT within 90 days, or cell therapy within 90 days of start of therapy;
* History of Grade ≥ 3 CRS or Grade ≥ 3 ICANS;
* Active and uncontrolled infections;
* Unresolved AEs ≥2 Grade due to prior anticancer therapies, with some exceptions

The above is a summary, other exclusion criteria details may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-02-14 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicities (DLTs). | Module 1 - From the first administration of AZD5492 until the end of cycle 1 (up to 5 weeks).
  DLTs are dose-limiting toxicities as defined in the study protocol.
Safety evaluation of AZD5492: Number of participants with treatment-related adverse events. | Module 1 - From the first administration of AZD5492 within the duration of the treatment period, up to and including 90 (+7) days after the last dose of study treatment , but prior to subsequent cancer therapy.
  Incidence and severity of AEs, AESIs, and SAEs
Tolerability evaluation of AZD5492: Number of participants with treatment-related adverse events. | Module 1 - From the first administration of AZD5492 within the duration of the treatment period, up to and including 90 (+7) days after the last dose of study treatment , but prior to subsequent cancer therapy.
  SAEs/AEs leading to discontinuation of AZD5492.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Module 1 - From first dose of AZD5492 up to 2 years after last dose.
  The proportion of participants with a complete response or partial response, according to Lugano criteria for malignant lymphoma and iwCLL 2018 criteria for CLL.
Complete Response Rate (CR Rate) | Module 1 - From first dose of AZD5492 up to 2 years after last dose.
  The proportion of participants with a complete response (CR), according to Lugano criteria for malignant lymphoma and iwCLL 2018 criteria for CLL.
Duration of Response (DoR) | Module 1 - From first dose of AZD5492 up to 2 years after last dose.
  The time from the date of first documented response until the date of documented progression (according to Lugano criteria for malignant lymphoma and iwCLL 2018 criteria for CLL) or death due to any cause.
Progression-free Survival (PFS) | Module 1 - From first dose of AZD5492 up to 2 years after last dose.
  The time from the date of first dose until the date of documented disease progression (according to Lugano criteria for malignant lymphoma and iwCLL 2018 criteria for CLL) or death due to any cause.
Overall Survival (OS) | Module 1 - From first dose of AZD5492 up to 2 years after last dose.
  The time from the date of first dose until date of death due to any cause.
Pharmacokinetics of AZD5492: serum concentration of study drug | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  Maximum observed serum concentration of AZD5492.
Pharmacokinetics of AZD5492: Maximum plasma concentration of the study drug (Cmax). | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  Maximum observed plasma concentration of AZD5492.
Pharmacokinetics of AZD5492: Area under the concentration time curve (AUC). | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  Area under the plasma concentration-time curve.
Pharmacokinetics of AZD5492: apparent clearance | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  The volume of plasma from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD5492: Half-life (t 1/2) | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  Terminal elimination half-life.
To determine the immunogenicity of AZD5492 | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  The number of participants who develop ADAs measured in serum.
To determine the immunogenicity of AZD5492 | Module 1 - From informed consent until 90 days after last dose of AZD5492.
  The percentage of participants who develop ADAs measured in serum.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (8):
  - Research Site, La Jolla, California
  - Research Site, Boston, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Nedlands
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (2):
  - Research Site, Hangzhou
  - Research Site, Shanghai
- Research Site, København Ø, Denmark
- France (2):
  - Research Site, Pessac
  - Research Site, Villejuif
- Germany (3):
  - Research Site, München
  - Research Site, Ulm
  - Research Site, Würzburg
- Italy (2):
  - Research Site, Bologna
  - Research Site, Milan
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa
- Spain (3):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://www.astrazenecaclinicaltrials.com/our-transparency-commitments/.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://www.astrazenecaclinicaltrials.com/our-transparency-commitments/.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://www.vivli.org